CLINICAL TRIAL: NCT06759571
Title: Impact of Photobiomodulation Bone Healing Following Cystic Enucleation: A Randomized Clinical Trial
Brief Title: Impact of Photobiomodulation Bone Healing Following Cystic Enucleation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Tarek Abdelbarry, Lecturer of Oral and Maxillofacial Surgery, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Photobiomodulation
Record Dates: First submitted 2024-12-28; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-02

CONDITIONS: Maxillary Cyst

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): About 10 patients who will be subjected to low intensity diode laser "soft-laser SL202" ("PERTO LASER", pr. Stachek, 47, Saint Petersburg, Russia) before surgery (two times / week for two weeks) and then following surgery (for three times per week for four weeks).
  Interventions: Procedure: low level laser treatment
- Group B (Active Comparator): About 10 patients who will undergo conventional surgical enucleation of intra-body maxillary cystic lesions.
  Interventions: Procedure: low level laser treatment

INTERVENTIONS:
Procedure: low level laser treatment — to evaluate the effect of low-level laser therapy (LLLT) bone healing when used prior and following enucleation of intra-body maxillary cystic lesions
  Other Names: Maxillary cystic enucleation

SUMMARY:
A well-known issues confronted by oral and maxillofacial specialists are the osseous defects and dead spaces and how can be obliterated and augmented in the facial regions. Unerupted tooth and bone loss after its removal, remaining roots and enucleation of cysts; all of which makes prosthetic rehabilitation and implant application more complicated

DETAILED DESCRIPTION:
Bone is undergoes remodeling via cycles of bone resorption and bone formation which is considered a mineralized connective tissue, an inflammatory immune reaction which is triggered by local injury which is thought to highly influence the outcome of the bone healing process.

Low-Level Laser Therapy (LLLT) is a form of phototherapy that involves the application of low power monochromatic and coherent light to areas of injuries and lesions. It has been shown to induce wound healing in non-healing bone defects .

Bone healing is a multidimensional process of reconstruction of the bone tissue with an overlapping timeline. Because of the regeneration ability of the bone, bone defects can heal spontaneously under suitable physiological environmental conditions. The healing process of the bone defect is time consuming, and new bone generation takes place slowly because of diminished of blood supply to the defect site and insufficiency of calcium and phosphorus to strengthen and harden new bone.

The low-level laser therapy (LLLT) has a positive effect on bone tissue metabolism . Moreover it is beneficial for the initial stages of alveolar bone healing and for further calcification; An experimental animal study in both diabetic and normal rats under histological observations and gene expression analyses have confirmed this when applied at a dose of 13.95 J/cm2 for 60 sec .

ELIGIBILITY:
Inclusion Criteria:

- patients (class I category according to American society of anesthesiologists) over 20 years and under 50 years of age, of either gender who are seeking cyst enucleation of painful intra-body maxillary cystic lesions 3 x 4 cm in size.

Exclusion Criteria:

* any systemic disease that interferes with bone healing,
* patients with significant medical condition,
* alcoholic individuals,
* patients on drugs that affect the central nervous systems,
* patients who reported the use of drugs that might interfere with pain sensitivity
* pregnancy,
* lactation

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Post- operative pain assessment | From First 24 hours after The procedure till 7 days
  Pain scores will be recorded on visual analog scale (VAS) using a 0 to 10 pain score basis with 0 being no pain and 10 being the worst pain the patient had ever experienced.(record will be every 24h for 7 days)

SECONDARY OUTCOMES:
Radiographic assessment | From baseline to 3 and 6 months after the operation day
  CBCT (Planmeca. Promax 3DMid machine, Helsinki Finland) scan will be obtained immediately post-operative, 3 and 6 months postoperative.

CONTACTS AND LOCATIONS:
Overall Officials: TAREK ABDELBARY, Lecturer, Principal Investigator — Faculty of Dentistry, Minia University
Locations (1):
- Faculty of Dentistry, Minia University, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided